CLINICAL TRIAL: NCT05740605
Title: Implementation of a HABIT-ILE at Home Intervention for Children With Bilateral Cerebral Palsy: a Non-inferiority Randomized Controlled Trial
Brief Title: Implementation of a HABIT-ILE Intervention at Home for Children With Bilateral Cerebral Palsy
Acronym: HABITILEhome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B4032022000142a
Record Dates: First submitted 2023-02-02; First posted 2023-02-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: HABIT-ILE; Intensive therapy based on motor skill learning; Home rehabilitation; Caregiver; Telerehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The trial will be a single-blind, randomized, monocentric controlled trial. The trial start with a division in two arms HABIT-ILE therapy classic or at home then half of each group will benefit from a HABIT-ILE follow-up while the other will have usual care. That means that participants will be divided into four groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary aim, the GMFM, will be videotaped and the scoring will be done by a blind evaluator. In secondary outcomes, the BoHA will be blind scored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HABIT-ILE therapy at home without a HABIT-ILE follow-up at home (Experimental): 2 weeks of HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) therapy at home followed by 9 weeks of usual care
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities at home; Behavioral: Usual Care
- HABIT-ILE therapy at home with a HABIT-ILE follow-up at home (Experimental): 2 weeks of HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) therapy at home followed by 9 weeks of HABIT-ILE follow-up at home
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities at home; Behavioral: Follow-up Hand-Arm Bimanual Intensive Therapy Including Lower Extremities
- Classic HABIT-ILE therapy without follow-up HABIT-ILE at home (Active Comparator): 2 weeks of classic HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) therapy on site followed by 9 weeks of usual care
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE); Behavioral: Usual Care
- Classic HABIT-ILE therapy with follow-up HABIT-ILE at home (Active Comparator): 2 weeks of classic HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) therapy on site followed by 9 weeks of HABIT-ILE follow-up at home
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE); Behavioral: Follow-up Hand-Arm Bimanual Intensive Therapy Including Lower Extremities

INTERVENTIONS:
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) — HABIT-ILE ("Hand-Arm Bimanual Intensive Therapy including Lower Extremities") is an intensive therapy that continuously incorporates postural control and LE function. This motor learning-based approach include specificity of the practice, motivation, shaping of the task, intensive blocks of training and Hands-Off. Moreover, the therapy is goal-oriented to increase functional independence during daily living. This therapy has shown impressive improvements in children with PC.
  Arms: Classic HABIT-ILE therapy with follow-up HABIT-ILE at home; Classic HABIT-ILE therapy without follow-up HABIT-ILE at home
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities at home — The HABIT-ILE therapy at home will follow the same principles as the classic HABIT-ILE. The therapy will take place in the patient's home and a close person (caregiver) will accompany the patient during the therapy. A device will be used to facilitate the implementation of home therapy. Supervision of the therapeutic process will be done remotely by a team of trained supervisors. One hour of remote supervision per day will be scheduled within 6.5 hours of therapy.
  Other Names: HABIT-ILE@home
  Arms: HABIT-ILE therapy at home with a HABIT-ILE follow-up at home; HABIT-ILE therapy at home without a HABIT-ILE follow-up at home
Behavioral: Follow-up Hand-Arm Bimanual Intensive Therapy Including Lower Extremities — HABIT-ILE follow-up at home follow the same principles as classic HABIT-ILE but is delivered at the patient home with 4 hours per week in autonomy and 1 hour per week under supervision.
  Other Names: Follow-up HABIT-ILE@home
  Arms: Classic HABIT-ILE therapy with follow-up HABIT-ILE at home; HABIT-ILE therapy at home with a HABIT-ILE follow-up at home
Behavioral: Usual Care — Usual care is all the weekly physiotherapy and occupational therapy sessions that the patient usually receives.
  Other Names: Customary care
  Arms: Classic HABIT-ILE therapy without follow-up HABIT-ILE at home; HABIT-ILE therapy at home without a HABIT-ILE follow-up at home

SUMMARY:
Intensive interventions based on the principles of motor skill learning, like Hand-Arm Bimanual Therapy Including Lower Extremities (HABIT-ILE), have demonstrated excellent effectiveness in improving motor function and daily life independence of children with cerebral palsy (CP). Patients living far from big cities do not have easy access to such interventions, usually applied in the form of camps. This randomized controlled trial will include 48 children with bilateral CP and aims to test a home version of HABIT-ILE with the use of a specifically designed virtual device and a remote supervision. For this purpose, two types of two weeks intensive treatment programs will be compared: Hand and Arm Bimanual Intensive Therapy Including Lower Extremities at home ("HABIT-ILE at home") and "classic HABIT-ILE". Moreover, this study also aims to assess whether the patient's abilities are better with a follow-up at home after two weeks of HABIT-ILE therapy than without follow-up post therapy. Four groups will be compared: HABIT-ILE at home therapy with a follow-up at home, HABIT-ILE at home therapy without follow-up, classic HABIT-ILE therapy with a follow-up at home and classic HABIT-ILE therapy without follow-up. Children will be assessed at 3 time points: before therapy, after therapy and 3 months after the start of therapy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common cause of physical disability in children: it occurs in 1 to nearly 4 children in 1000 newborns worldwide. This major public health issue caused by abnormal brain development or damage during brain development result in different symptoms that vary from one patient to another. Even if all children with CP will develop motor symptoms (abnormal movement patterns and posture) some of them will also develop non-motor symptoms such as pain (75%), intellectual deficits (50%), language disorders (25%), epilepsy (25%), behavioral and sleep disorders (20-25%). The consequences of these symptoms are very variable and result in long-term functional deficits in the activities of daily living, such as dressing, eating, going to the bathroom, etc. To improve these patients' autonomy, intensive therapies based on motor skill learning (MSL) have been shown to be especially effective. Among these therapies, Hand-Arm Bimanual Intensive Therapy including Lower Extremities (HABIT-ILE) has been developed over the last decade in the MSL-IN laboratory of UCLouvain and has shown impressive improvements in children with CP. It is based on an intensive training of bimanual activities, with a systematic inclusion of lower limbs and trunk motor control. This therapy is given in the form of a rehabilitation camp of at least 50 hours on site. Therefore, the implementation of a classic HABIT-ILE, in day-camp requires a great commitment from the families who must travel to the camp location for two weeks of therapy. In addition, for patients living far from big cities or unable to travel, access to these therapies can be really complex. Moreover, these camps are applied in a group of 8-12 children. Each participant is accompanied by at least one therapist (physiotherapist or occupational therapist and sometimes student) trained in HABIT-ILE therapy. This implies that a HABIT-ILE camp requires minimum 12 trained therapists. Nonetheless, there is a lack of therapists that makes the implementation of these camps still challenging. In addition, the health requirements related to COVID-19 make it difficult to implement any kind of therapy and to assess patients' progress. Therefore, this health crisis has highlighted the importance of being able to offer home-based therapy. To answer the problematics of pandemic, accessibility and of lack of HABIT-ILE therapists, the idea of implementing HABIT-ILE at home was born. How could we implement MSL principles at home? Some of the key components of MSL are intensity, shaping of the task (with part- task and increasing difficulty), goal-oriented therapy, positive reinforcement and hands-off (voluntary movements by the patients, not guided by the therapist). To incorporate those principles and ensure the validity of the therapy, guidance by a trained HABIT-ILE supervisor is necessary. This supervision will be provided through remote telerehabilitation sessions. Virtual reality is well suited to implement MSL-IN principles and allows for remote communication with patients. Tele-reeducation devices are numerous: from classic commercials video game found in stores to devices made for rehabilitation. Alone these devices do not allow the implementation of all the principles of motor skill learning but with the supervision of therapists trained in HABIT-ILE supervision, this objective could be achieved. With the help of new technologies, will the HABIT-ILE supervisors be able to implement HABIT-ILE at home in a reliable and standardized way for children with CP aged 6 to 18 ? This RCT aims to assess if HABIT-ILE at home is not inferior to HABIT-ILE in camp regarding physical abilities, functional activities and participation of the participants.

Moreover, if the maintenance of skills during HABT-ILE camp at 3- and 6-months post-therapy has been proven, the question of improving them has not been investigated yet. Indeed, we know that in order to maintain the skills learned during the HABIT-ILE therapy, it is necessary to practice them on a daily basis. If a skill is not used it will lead to a cortical reorganization of the motor cortex at the expense of this skill. Thus, there is a persistent cycle of decreased utilization that leads to unfavorable cortical reorganization that leads to decreased utilization, etc. It is called "learned non-use". In order to reduce this phenomenon and thus improve the transfer of the HABIT-ILE skills into the daily life of the children, we wonder about the benefit of a post-therapy follow-up. Once again, the use of tele-rehabilitation can provide us a solution of daily delocalized therapy directly implemented at the patient's home and supervised remotely. Could the transfer of learned skills be improved with a follow-up at home post therapy? In order to answer this question, after the two weeks of both HABIT-IL modality, we will set up a HABIT-ILE telerehabilitation follow-up for 9 weeks. This study therefore also aims to assess if the patient's abilities could be potentialize with a follow-up than without a follow-up after two weeks of HABIT-ILE therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed diagnosis of bilateral Cerebral Palsy
* Age 5 to 18 years old
* Ability to interact and understand simple instructions in order to complete assessments and therapy
* Availability of a caregiver for 6h30 per day during two weeks of therapy

Exclusion Criteria:

* Uncontrolled seizure
* Botulinum toxin injection in the last 6 months before the first assessment or during the therapy
* Intensive therapy in the last 6 months before the first assessment or during the therapy
* Surgery that could affect the assessments or therapy in the last 6 months before the first assessment or during the therapy
* Severe visual or cognitive impairments interfering with treatment and or assessments
* Any typical contraindication for MRI

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change on Gross Motor Function (GMFM-66) | baseline, 2 weeks and 12 weeks after baseline
  Developed to assess the changes in gross motor function of children with cerebral palsy (scored in percentage)

SECONDARY OUTCOMES:
Changes in the Both Hand Assessment (BOHA) | baseline, 2 weeks and 12 weeks after baseline
  The BoHA aims to measure the effective use of both hands in bimanual activity performance, as well as to quantify the possible side difference between hands. (score in percentage)
Changes in gross unimanual dexterity by the Box and block test (BBT) | baseline, 2 weeks and 12 weeks after baseline
  The BBT assess unimanual dexterity by quantifying the maximum of wooden blocks transferred from one space to the other during 1 minute (Higher scores indicate better performance)
Changes in the Six Minutes' Walk Test (6MWT) | baseline, 2 weeks and 12 weeks after baseline
  The 6MWT assess endurance while walking 6 minutes without pause. More distance walked (in meters) indicate better performance
Changes in activities of daily living assessed by ABILHAND-Kids questionnaires. | baseline, 2 weeks and 12 weeks after baseline
  ABILHAND-Kids is a questionnaire that measures manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. ABILHAND-Kids has been validated in cerebral palsy children (age 6-15). 21 manual activities perceived by the children parents. Each item is answered on a 3-level scale (impossible, difficult, easy). The item difficulty increases with bimanual involvement: higher score means better performance
Changes in activities of daily living assessed by PEDI questionnaire | baseline, 2 weeks and 12 weeks after baseline
  This parent's filled questionnaire measures the performance of the child in the daily life activities and movement domains, focusing on the capacity of upper extremities and lower extremities during these activities. It ranges from 0 to 100% (higher score means better performance)
Changes in activities of daily living assessed by ACTIVLIM-CP Questionnaire | baseline, 2 weeks and 12 weeks after baseline
  This parent's filled questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower extremities through 43 items specific to patients with cerebral palsy. It ranges from - 7 to +7 logits (higher score means better performance)
Changes in activities of locomotion assessed by ABILOCO-Kids Questionnaire | baseline, 2 weeks and 12 weeks after baseline
  The ABILOCO-Kids questionnaire is a measure of locomotion ability for children with lower limb impairments. The scale has been calibrated in children with cerebral palsy (age 6-15). The Parent is asked to fill in the questionnaire by estimating their child's ease or difficulty in performing each activity. During the evaluation, the 3-level response scale is presented to the parent. The parent is asked to rate his/her perception on the response scale as 'Impossible', 'Difficult' or 'Easy'. The activities not attempted by the child within the last 3 months are not scored and are entered as not applicable (check the question mark '?' on the scoring sheet). The activities that the child does not perform because they are too difficult must be scored as 'Impossible'. (higher score means better performance)
Changes in the fine motor skills and functional activities of the hand assessed by the Jebsen Hand Fuction Test | baseline, 2 weeks and 12 weeks after baseline
  The Jebsen Hand Function Test (JHFT) assesses fine motor skills, weighted and non-weighted hand function activities during performance of activities of daily living. The JHFT consists of 6 items that measure: (a) fine motor skills; (b) weighted functional tasks; and (c) non-weighted functional tasks:
  Turning over a 3×5-inch card Picking up small common objects Simulated feeding Stacking checkers Picking up large light cans Picking up large heavy cans
Changes in self-esteem assessed by the ESTIMILL-CP questionnaire | baseline, 2 weeks and 12 weeks after baseline
  The ESTIMILL-CP is self-completed by the children. It consists of 26 illustrated items where the child must choose between "I identify with the situation" or "I don't identify with the situation" and then whether it's "a lot of similarity" or "not much". The lower the score, the worse the self-esteem.
Changes in the PILS-CP questionnaire. | baseline, 2 weeks and 12 weeks after baseline
  The PILS-CP questionnaire self-administrated (patients do not realize the life situation). Patients are asked to estimate the involvement in performing each life situation. During the evaluation, a 3-level response scale is presented to the patients. Patients are asked to rate their participation on the response scale as either "I am not involved", "I am a little bit involved", "I am fully involved". Life situations that the patients do not want to be involve are rated with "?"
Changes in lower limbs physical activity | During the 2 weeks of therapy
  With a movement sensor on each wrist and on the leg, the percentage of total time spent in movement (Standing, walking or sitting) is measured. Calculated in terms of the changes in the acceleration (m/s²).
Changes in upper limbs physical activity | During the 2 weeks of therapy
  With a movement sensor on each wrist and on the leg, the activities of both hand is quantified. Calculated in terms of the changes in the acceleration (m/s²).
Changes in the functional goals assessed by the Canadian Occupational Performance Measure (COPM) questionnaire. | baseline, 2 weeks and 12 weeks after baseline
  In this interview, patients set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the patient's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10)
Changes in 3D T1-weighted structural imaging. | baseline, 2 weeks and 12 weeks after baseline
  This sequence allows to measure changes in gray matter (cortical thickness)
Changes on the Fractional Anisotropy (Diffusion tensor imaging (DTI)) | baseline, 2 weeks and 12 weeks after baseline
  This sequence allows to measure changes in the fractional anisotropy (FA) on the white matter tracts. FA is a scalar value (no unit) between zero and one that describes the degree of anisotropy of white matter water molecules.
Changes on RS-fMRI | baseline, 2 weeks and 12 weeks after baseline
  Resting-state functional magnetic resonance imaging (rs-fMRI) evaluates the regional interactions that occur during the resting or task-negative state. The magnitude of the brain activation during rs-fMRI will be assessed
Changes on the Mean Diffusivity (Diffusion tensor imaging (DTI)) | baseline, 2 weeks and 12 weeks after baseline
  This sequence allows to measure the mean changes in the diffusivity (MD). MD is a scalar value (no unit) between zero and one that describes the degree of molecular diffusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, Phd, Prof., Principal Investigator — Université Catholique de Louvain
Locations (1):
- MSL-IN Lab, Institue of Neurosciences, UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Sakzewski L, Bleyenheuft Y, Boyd RN, Novak I, Elliott C, Reedman S, Morgan C, Pannek K, Fripp J, Golland P, Rowell D, Chatfield M, Ware RS. Protocol for a multisite randomised trial of Hand-Arm Bimanual Intensive Training Including Lower Extremity training for children with bilateral cerebral palsy: HABIT-ILE Australia. BMJ Open. 2019 Sep 8;9(9):e032194. doi: 10.1136/bmjopen-2019-032194. PMID 31501133
- [Background] Bleyenheuft Y, Gordon AM. Hand-arm bimanual intensive therapy including lower extremities (HABIT-ILE) for children with cerebral palsy. Phys Occup Ther Pediatr. 2014 Nov;34(4):390-403. doi: 10.3109/01942638.2014.932884. Epub 2014 Oct 1. PMID 25271469
- [Background] Demers M, Fung K, Subramanian SK, Lemay M, Robert MT. Integration of Motor Learning Principles Into Virtual Reality Interventions for Individuals With Cerebral Palsy: Systematic Review. JMIR Serious Games. 2021 Apr 7;9(2):e23822. doi: 10.2196/23822. PMID 33825690
- [Background] Bleyenheuft Y, Dricot L, Gilis N, Kuo HC, Grandin C, Bleyenheuft C, Gordon AM, Friel KM. Capturing neuroplastic changes after bimanual intensive rehabilitation in children with unilateral spastic cerebral palsy: A combined DTI, TMS and fMRI pilot study. Res Dev Disabil. 2015 Aug-Sep;43-44:136-49. doi: 10.1016/j.ridd.2015.06.014. Epub 2015 Jul 13. PMID 26183338